CLINICAL TRIAL: NCT06606210
Title: An Observer-Blinded Multicenter Randomized Controlled Trial Evaluating Porcine Placental Extracellular Matrix as an Adjunct to Standard of Care Versus Standard of Care Alone in Hard-to-Heal Venous Leg Ulcers
Brief Title: INNOVEN: Efficacy of Porcine Placental Extracellular Matrix Plus Standard of Care (SOC) Versus SOC Alone
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ConvaTec Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WC-24-454
Record Dates: First submitted 2024-09-13; First posted 2024-09-20 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Wound Heal; Venous Leg Ulcer
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard of Care (No Intervention): Compression, debridement, reduction of bacterial burden, and proper moisture balance.
- Standard of Care plus Interventional Device (Experimental): Weekly applications of the study device in conjunction with standard of care including compression, debridement, reduction of bacterial burden, and proper moisture balance,
  Interventions: Device: InnovaMatrix® AC

INTERVENTIONS:
Device: InnovaMatrix® AC — Weekly dressing applications
  Other Names: Porcine Derived Extracellular Matrix
  Arms: Standard of Care plus Interventional Device

SUMMARY:
INNOVEN is a multi-center randomized controlled clinical trial to evaluate the efficacy of porcine placental extracellular matrix (PPECM) and standard of care (SOC) versus SOC alone in the closure of non-healing venous leg ulcers (VLUs).

DETAILED DESCRIPTION:
An Observer-Blinded Multicenter Randomized Controlled Trial Evaluating Porcine Placental Extracellular Matrix as an Adjunct to Standard of Care versus Standard of Care Alone in Hard-to-Heal Venous Leg Ulcers.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be at least 21 years of age or older.
2. At randomization subjects must have a target ulcer with a minimum surface area of 1 cm2 and a maximum surface area of 25 cm2 measured post-debridement.
3. The target ulcer must have been present for a minimum of 4 weeks and cannot have received more than 52 weeks of high-level compression prior to the initial screening visit.
4. No visible signs of improvement in the four weeks prior to randomization: less than 40% reduction in wound size over the 4 weeks prior to randomization.
5. The affected limb must have adequate perfusion confirmed by vascular assessment. Any of the following methods performed within 3 months of the first screening visit are acceptable:

   1. ABI between 0.7 and ≤ 1.3;
   2. TBI ≥ 0.6;
   3. TCOM ≥ 40 mmHg;
   4. PVR: biphasic.
6. If the potential subject has two or more ulcers, they must be separated by at least 2 cm post-debridement. The largest ulcer satisfying the inclusion and exclusion criteria will be designated as the target ulcer.
7. The potential subject must agree to attend the weekly study visits required by the protocol.
8. The potential subject must be willing and able to participate in the informed consent process.

Exclusion Criteria:

1. The potential subject is known to have a life expectancy of < 6 months.
2. The target ulcer exhibits signs or symptoms consistent with clinical infection, requiring topical antibiotic or antimicrobial agents or systemic antibiotic therapy, or there is cellulitis in the surrounding skin.
3. The target ulcer exposes tendon or bone.
4. There is evidence of osteomyelitis complicating the target ulcer.
5. The potential subject is receiving immunosuppressants (including systemic corticosteroids at doses greater than 10 mg of prednisone per day or equivalent) or cytotoxic chemotherapy or is taking medications that the Principal Investigator believes will interfere with wound healing (e.g., biologics).
6. The potential subject has applied topical steroids to the ulcer surface within one month of initial screening.
7. The potential subject has glycated hemoglobin (HbA1c) greater than or equal to 12% within 3 months of the initial screening visit.
8. The surface area of the target ulcer has reduced in size by more than 20% in the 2 weeks prior to the initial screening visit ("historical" run-in period). Digital planimetry is not required for measurements taken during the historical run-in period (e.g., calculating surface area using length X width is acceptable).
9. The surface area measurement of the target ulcer decreases by 20% or more during the active 2-week screening phase: the 2 weeks from the initial screening visit (SV-1) to the TV-1 visit during which time the potential subject received SOC.
10. The potential subject has had a lower extremity Deep Vein Thrombosis (DVT) to either limb within the previous 90 days.
11. The potential subject is unable to tolerate therapeutic compression (30-40mmHg).
12. Women who are pregnant or considering becoming pregnant within the next 6 months.
13. The potential subject has end stage renal disease requiring dialysis.
14. Participation in another clinical trial involving treatment with an investigational product within the previous 30 days.
15. A potential subject who, in the opinion of the Investigator, has a medical or psychological condition that may interfere with study assessments.
16. The potential subject was treated with hyperbaric oxygen therapy (HBOT) or a Cellular, Acellular, Matrix-like Product (CAMP) in the 30 days prior to the initial screening visit.
17. The potential subject has a malnutrition indicator score <17 as measured on the Mini Nutritional Assessment.
18. Potential subjects with a sensitivity or allergy to porcine materials or collagen.
19. Potential subjects with religious or personal objection to use of porcine- or animal-derived materials.
20. A subject with a disorder that would create unacceptable risk of treatment complications.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-09-19 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Determine the efficacy of Porcine Placental Extracellular Matrix (PPECM) plus Standard of Care (SOC) versus SOC alone in achieving complete closure of hard-to-heal venous leg ulcers over 12 weeks. | 12 weeks
  The percentage of target ulcers achieving complete wound closure defined as complete epithelialisation of the wound surface.

SECONDARY OUTCOMES:
Determine the time to closure for ulcers achieving complete closure over 12-weeks for PPECM+SOC versus SOC alone. | 12 weeks
  For study ulcers achieving complete closure, the time to closure over the 12-week treatment duration.
Determine the percent area reduction (PAR) of the ulcer over the 12-week treatment period. | 12 weeks
  Percentage wound area reduction from initial treatment to 12-week measured weekly with digital photographic planimetry.
Determine quality of life (QoL) for subjects receiving PPECM+SOC compared to SOC alone. | Day 0, 4 weeks, 8 weeks, and 12 weeks
  Measured with Forgotten Wound Score (FWS) questionnaire, assessing the awareness of the wound, ranging from "Never" to "Mostly").
Determine quality of life (QoL) for subjects receiving PPECM+SOC compared to SOC alone. | Day 0, 4 weeks, 8 weeks, and 12 weeks
  Measured with standard Wound Quality of Life (wQOL) questionnaire, assessing how wound care has affected the quality of life in the last seven days, ranging from "Not at all" to "Very much".
Determine the long-term durability of closure in PPECM+SOC versus SOC alone. | 3-, 6-, 9-, and 12-months after wound closure or completion of the initial 12-week treatment phase
  Change in quality of life using the Wound Quality of Life (wQOL) questionnaire, assessing how wound care has affected the quality of life in the last seven days, ranging from "Not at all" to "Very much".
Determine the long-term durability of closure in PPECM+SOC versus SOC alone. | 3-, 6-, 9-, and 12-months after wound closure or completion of the initial 12-week treatment phase
  Change in quality of life using the Forgotten Wound Score (FWS) questionnaire, assessing the awareness of the wound, ranging from "Never" to "Mostly").

OTHER OUTCOMES:
Number of serious adverse events (SAE). | 12 month
  Number of events related to the device, procedure, or target study ulcer.
Number of study-ulcer infections. | 12 month
  Infections for PPECM+SOC vs SOC alone.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E. Serena, MD FACS, Principal Investigator — SerenaGroup, Inc.
Locations (1):
- Three Rivers Wound and Hyperbaric Center, North Port, Florida, United States

IPD SHARING:
Plan to Share IPD: No